CLINICAL TRIAL: NCT03274648
Title: Therapeutic Modulation of Butyrate Production in Behçet's Patients: a Dietary Intervention Trial
Brief Title: Dietary Interventions and Butyrate Production in Behçet's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, GIACOMO EMMI, Principal Investigator, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: butyrate2017
Record Dates: First submitted 2017-08-31; First posted 2017-09-07 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Behcet Syndrome
MeSH Terms: conditions — Behcet Syndrome | interventions — Butyrates; Diet, Vegetarian

STUDY DESIGN:
Intervention Model Description: Behçet's will be assigned to one of the following treatments:
  * vegetarian diet containing inulin and resistant starch-rich foods, including no meat and fish, but containing eggs and dairy products
  * habitual diet supplemented with 2.4g/day of oral butyrate
  * habitual diet without supplementation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- vegetarian diet (Experimental): vegetarian diet containing inulin and resistant starch-rich foods, including no meat and fish, but containing eggs and dairy products
  Interventions: Dietary Supplement: Vegetarian diet
- Habitual diet + oral butyrate (Experimental): habitual diet supplemented with 2.4g/day of oral butyrate
  Interventions: Dietary Supplement: Oral butyrate
- Habitual diet (Active Comparator): habitual diet without supplementation
  Interventions: Dietary Supplement: Habitual diet

INTERVENTIONS:
Dietary Supplement: Oral butyrate — Patients follow the habitual diet supplemented with 2.4g/day of oral butyrate
  Arms: Habitual diet + oral butyrate
Dietary Supplement: Vegetarian diet — Patients follow a vegetarian diet containing inulin and resistant starch-rich foods, including no meat and fish, but containing eggs and dairy products
  Arms: vegetarian diet
Dietary Supplement: Habitual diet — Patients follow the habitual diet
  Arms: Habitual diet

SUMMARY:
A dietary intervention trial will be performed on patients affected by Behçet's syndrome. Three different diets will be compared, analyzing their effects on the gut microbiota composition, on endogenous butyrate production and on the general symptoms in Behçet's patients.

DETAILED DESCRIPTION:
A dietary intervention trial will be conducted with the use of three different diets in order to compare the effects of these diets on the gut microbiota composition, on endogenous butyrate production and on the general symptoms in Behçet's patients.

The study will be a randomized, open trial designed to test whether a vegetarian diet or an habitual diet supplemented with oral butyrate would benefit the butyrate production, the gut microbiota composition and the general symptoms of Behçet's patients, compared with the habitual diet.

The study will involve 30 subjects with Behçet syndrome. Patients will be randomly assigned to follow a 3-months isocaloric dietary profile with either:

* vegetarian diet containing inulin and resistant starch-rich foods, including no meat and fish, but containing eggs and dairy products
* habitual diet supplemented with 2.4g/day of oral butyrate
* habitual diet without supplementation At the baseline visit, subjects will be educated about the aims and methods of the clinical trial and will sign their informed consent form.

Anthropometric measurements, body composition, and blood and stool sampling will be obtained from each participant at the beginning and at the end of the intervention period. All subjects will be examined between 07.00 and 09.30 hours after a 12 h fasting period.

The following parameters will be analyzed both at the beginning and at the end of the intervention period:

* Complete blood count
* Lipid variables - total cholesterol, low density lipoprotein cholesterol (LDL), high density lipoprotein cholesterol (HDL), triglycerides
* Glycemic profile - glucose, insulin, glycated hemoglobin (HbA1C), HOMA index
* Liver function tests - aspartate aminotransferase (AST), alanine transaminase (ALT), gammaglutamyl transferase (GGT), alkaline phosphatase (ALP), albumin, prealbumin
* Kidney function tests - serum creatinine, urea, uric acid
* Mineral profile - sodium, potassium, magnesium, calcium
* Iron metabolism - iron, ferritin
* Vitamin profile - vitamin B12, folic acid, vitamin D
* Thyroid function - TSH
* Inflammatory markers - erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), fibrinogen, serum amyloid A (SAA)
* Serology for celiac disease - IgA, anti-transglutaminase antibodies (IgA), anti endomysium antibodies (IgA)
* Circulating levels of inflammatory cytokines
* Oxidative stress markers
* Gut microbiota composition
* Butyrate production

At the beginning and at the end of the intervention period, participants will be asked to complete a questionnaire, which will assess Behçet's symptoms frequency and severity. In addition, participants will be contacted by phone to complete a 24-hours recall in order to test the adherence to diets they have been assigned to.

ELIGIBILITY:
Inclusion Criteria:

* All patients affected by Behçet's disease

Exclusion Criteria:

* Pregnancy or breastfeeding
* Presence of diabetes mellitus
* Presence of other immune-mediated diseases
* Presence or history of cancer in the last 5 years
* Presence of infectious diseases in the last 3 months
* No antibiotic therapy in the last 3 months
* No vegetarian or vegan diet
* No intake of pro- or pre-biotics in the last 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of gut microbiota composition | 0-3 months
Evaluation of butyrate production | 0-3 months
  For the extraction of SCFAs (and butyrate in particular) the method described in Schnorr et al. will be follow" [Schnorr SL, Candela M, Rampelli S, Centanni M, Consolandi C, Basaglia G,et al. Gut microbiome of the Hadza hunter-gatherers. Nat Commun 2014;5:3654]
Complete blood count | 0-3 months
  composite score
Lipid variables | 0-3 months
  composite score taking into account the levels of: total cholesterol, low density lipoprotein cholesterol (LDL), high density lipoprotein cholesterol (HDL), triglycerides
Glycemic profile | 0-3 months
  composite score taking into account the levels of : glucose, insulin, glycated hemoglobin (HbA1C), HOMA index
Vitamin profile | 0-3 months
  composite score, taking into account the levels of: vitamin B12, folic acid, vitamin D
Liver function tests | 0-3 months
  composite score taking into account the levels of: aspartate aminotransferase (AST), alanine transaminase (ALT), gammaglutamyl transferase (GGT), alkaline phosphatase (ALP), albumin, prealbumin
Kidney function tests | 0-3 months
  composite score taking into account the levels of : serum creatinine, urea, uric acid
Mineral profile | 0-3 months
  composite score taking into account the levels of: sodium, potassium, magnesium, calcium
Iron metabolism | 0-3 months
  composite score taking into account the levels of: iron, ferritin
Thyroid function | 0-3 months
  measurement of TSH levels
Inflammatory markers | 0-3 months
  composite score taking into account the levels of: erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), fibrinogen, serum amyloid A (SAA)
Serology for celiac disease | 0-3 months
  composite score taking into account the levels of: IgA, anti-transglutaminase antibodies (IgA), anti endomysium antibodies (IgA)
Circulating levels of inflammatory cytokines | 0-3 months
  composite score
Oxidative stress markers | 0-3 months
  composite score

SECONDARY OUTCOMES:
Evaluation Behçet's symptoms frequency and severity | 0-3 months
  Participants are asked to complete a questionnaire, which will assess Behçet's symptoms frequency and severity.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Background] Skef W, Hamilton MJ, Arayssi T. Gastrointestinal Behcet's disease: a review. World J Gastroenterol. 2015 Apr 7;21(13):3801-12. doi: 10.3748/wjg.v21.i13.3801. PMID 25852265
- [Background] Consolandi C, Turroni S, Emmi G, Severgnini M, Fiori J, Peano C, Biagi E, Grassi A, Rampelli S, Silvestri E, Centanni M, Cianchi F, Gotti R, Emmi L, Brigidi P, Bizzaro N, De Bellis G, Prisco D, Candela M, D'Elios MM. Behcet's syndrome patients exhibit specific microbiome signature. Autoimmun Rev. 2015 Apr;14(4):269-76. doi: 10.1016/j.autrev.2014.11.009. Epub 2014 Nov 27. PMID 25435420
- [Background] Wong JM. Gut microbiota and cardiometabolic outcomes: influence of dietary patterns and their associated components. Am J Clin Nutr. 2014 Jul;100 Suppl 1:369S-77S. doi: 10.3945/ajcn.113.071639. Epub 2014 Jun 4. PMID 24898225